CLINICAL TRIAL: NCT07163065
Title: Effect of Systemic Inflammatory Index and Other Biomarkers on Inferior Alveolar Nerve Block Success and Postoperative Pain
Brief Title: Evaluation of Systemic Inflammatory Index and Biomarkers in Relation to Inferior Alveolar Nerve Block Success and Postoperative Pain
Status: Active, not recruiting | Type: Observational
Sponsor: KEZBAN MELTEM ÇOLAK (Other)
Responsible Party: Sponsor-Investigator, KEZBAN MELTEM ÇOLAK, Professor of Endodontics, Principal Investigator, Ataturk University
Organization: Ataturk University (Other)
Other Study IDs: B.30.2.ATA.0.01.00/558
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain; Inferior Alveolar Nerve Block Failure; Inflammation Biomarkers; Dental Anesthesia Complications
Keywords: Systemic Inflammatory Index (SII); Neutrophil-to-Lymphocyte Ratio (NLR); Dental Anesthesia; Mandibular Block; Endodontic Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — Peripheral blood samples for hematological and inflammatory marker analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Undergoing Inferior Alveolar Nerve Block: Adult patients requiring dental treatment under inferior alveolar nerve block anesthesia. Participants will undergo standard IANB anesthesia, and postoperative pain will be evaluated along with systemic inflammatory markers obtained from blood samples.
  Interventions: Procedure: Inferior Alveolar Nerve Block Anesthesia

INTERVENTIONS:
Procedure: Inferior Alveolar Nerve Block Anesthesia — Standard inferior alveolar nerve block anesthesia performed with lidocaine and epinephrine for mandibular dental treatment. Success rate and postoperative pain outcomes will be recorded

SUMMARY:
This study aims to investigate the relationship between systemic inflammatory markers and the effectiveness of inferior alveolar nerve block anesthesia in patients undergoing dental treatment. The primary focus is on the Systemic Inflammatory Index (SII) and other inflammatory biomarkers, and how they may influence both the success of anesthesia and the intensity of postoperative pain. By analyzing blood samples and clinical outcomes, the study will provide new insights into the role of systemic inflammation in anesthesia effectiveness and postoperative pain control. The findings may help clinicians predict anesthetic success and improve pain management strategies in dental practice.

DETAILED DESCRIPTION:
Pulpitis is among the most common causes of orofacial pain. Irreversible pulpitis is characterized by a painful pulpal response to thermal stimuli that does not subside immediately after the removal of the stimulus. Pain is an unpleasant experience associated with actual or potential tissue damage. It is a subjective concept, and the pain threshold varies among individuals. Cold and heat tests are widely used in clinical practice for the diagnosis of symptomatic irreversible pulpitis. Irreversible pulpitis mainly arises due to infection caused by dental caries or the loss of restoration seal and microleakage. Dental trauma, pulpal exposure, and cracks can also lead to severe pulpitis. Pain associated with irreversible pulpitis accounts for more than 45% of emergency dental visits.

A detailed history of pain is essential, and it is often described as severe, dull, and throbbing; this pain may intensify with thermal or postural changes and can result in sleep disturbance. It tends to persist for prolonged periods (minutes to hours) and is generally unresponsive to analgesics. Patients also frequently report spontaneous and unprovoked sharp pains.

Achieving successful pulpal anesthesia during endodontic treatment of teeth with symptomatic irreversible pulpitis is critical for patient pain and stress management; however, this remains particularly challenging in mandibular teeth due to the inability of the inferior alveolar nerve block (IANB) to consistently provide profound anesthesia. Increased acidity in the inflamed pulp reduces the amount of basic anesthetic penetrating the nerve membrane, thereby delaying or preventing pulpal anesthesia.

Lip numbness, which typically occurs after anesthesia (i.e., loss of tactile sensation due to A-beta fiber blockade), is commonly regarded as an indicator that pulpal pain fibers (C and A-delta fibers) are also anesthetized and that the patient is ready for treatment. However, while tactile sensation is mediated by A-beta fibers, pain is transmitted via C and A-delta fibers. Local anesthetics block thick myelinated A-beta fibers and thin myelinated A-delta fibers at much lower concentrations than unmyelinated C fibers. Local anesthetics thus preferentially block myelinated fibers. Therefore, in healthy patients, the presence of lip numbness may be misleading for assessing pulpal anesthesia success. In patients with irreversible pulpitis, this method of assessment is even more unreliable.

**Several theories have been proposed to explain anesthetic failure. However, no studies have investigated the relationship between systemic inflammation and anesthetic success. The systemic immune-inflammation index (SII) is a novel biomarker for inflammation and is calculated as (neutrophil count × platelet count) / lymphocyte count. In our study, SII and other inflammatory markers will be evaluated. These additional inflammatory indices are as follows:

Aggregate index of systemic inflammation (AISI) = neutrophil count × monocyte count × platelet count / lymphocyte count

Platelet-to-lymphocyte ratio (PLR) = platelet count / lymphocyte count

Systemic inflammatory index (SII) = neutrophil count / PLR

Neutrophil-to-lymphocyte ratio (NLR) = neutrophil count / lymphocyte count.**

Moreover, although NLR has been used as an indicator of the inflammatory response in numerous diseases, there are insufficient data regarding its effects on postoperative pain, which is closely associated with acute inflammation. The aim of this study is to investigate the effects of systemic inflammatory markers, particularly SII and NLR, on the success of inferior alveolar nerve block anesthesia and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years.

Patients with a pain score greater than 54 on the Heft-Parker Visual Analog Scale (VAS).

Patients classified as ASA I according to the American Society of Anesthesiologists (ASA).

Teeth with probing depths less than 3 mm, suitable for rubber dam placement and restoration.

Vital mandibular molar teeth with a clinical diagnosis of irreversible pulpitis, confirmed by pulp vitality tests (electric pulp testing and cold testing).

Presence of bleeding upon access to the pulp chamber.

No use of non-steroidal anti-inflammatory drugs (NSAIDs) within the last 12 hours.

Absence of allergy to articaine.

Patient's consent to provide a blood sample.

Exclusion Criteria:

* Patients classified as ASA II or higher.

Pregnant women or those with suspected pregnancy.

Patients with periodontal pockets greater than 3 mm in the involved tooth.

Patients who received treatment with NSAIDs within the last 12 hours.

Patients allergic to articaine.

Teeth that had undergone previous endodontic treatment.

Teeth with extensive structural loss preventing rubber dam isolation.

Presence of internal or external root resorption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-65 years) requiring mandibular dental treatment under inferior alveolar nerve block anesthesia at Atatürk University Faculty of Dentistry, Department of Endodontics.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Success Rate of Inferior Alveolar Nerve Block Anesthesia | Within 15 minutes after injection
  Proportion of patients achieving successful anesthesia, defined as absence of pain during dental treatment following inferior alveolar nerve block.

CONTACTS AND LOCATIONS:
Overall Officials: KEZBAN MELTEM ÇOLAK, Principal Investigator — Atatürk University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Atatürk University Faculty of Dentistry, Department of Endodontics, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dziedzic EA, Gasior JS, Tuzimek A, Paleczny J, Junka A, Dabrowski M, Jankowski P. Investigation of the Associations of Novel Inflammatory Biomarkers-Systemic Inflammatory Index (SII) and Systemic Inflammatory Response Index (SIRI)-With the Severity of Coronary Artery Disease and Acute Coronary Syndrome Occurrence. Int J Mol Sci. 2022 Aug 23;23(17):9553. doi: 10.3390/ijms23179553. PMID 36076952
- [Background] Gibson PH, Croal BL, Cuthbertson BH, Small GR, Ifezulike AI, Gibson G, Jeffrey RR, Buchan KG, El-Shafei H, Hillis GS. Preoperative neutrophil-lymphocyte ratio and outcome from coronary artery bypass grafting. Am Heart J. 2007 Nov;154(5):995-1002. doi: 10.1016/j.ahj.2007.06.043. PMID 17967611
- See also: Related Info — https://www.aae.org